CLINICAL TRIAL: NCT04994145
Title: A Retrospective, Observational, Post-Market Clinical Investigation on Safety and Performance of Mepilex Border Post-Op for Post-Operative Wounds
Brief Title: A Post-Market Clinical Investigation on Mepilex Border Post-Op
Acronym: ARCTIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Other Study IDs: PD-612416
Record Dates: First submitted 2021-07-07; First posted 2021-08-06 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Surgical Wound
Keywords: Medical Device; Mepilex Border Post-Op; Knee replacement; Hip replacement; Surgical wound; Dressing; Wear time
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, observational (non-interventional), single-arm, single-centre, post-market clinical investigation designed to verify clinical performance and safety of Mepilex Border Post-Op when used according to clinical practice for post-operative wounds in a large and broad population.

The clinical investigation will consist of a retrospective medical record review, which will be completed with data from up to 450 female and male adult subjects who were treated with Mepilex Border Post-Op following elective hip or knee replacement at one clinic in Belgium between January 2016 and February 2021.

DETAILED DESCRIPTION:
Mepilex Border Post-Op is a CE-marked class IIa medical device developed, manufactured and marketed by Mölnlycke Health Care AB. This is a retrospective, observational (non-interventional), single-arm, single-centre, post-market clinical investigation designed to verify clinical performance and safety of Mepilex Border Post-Op when used according to clinical practice for post-operative wounds in a large and broad population. The overall objective of this investigation is to confirm the clinical performance of Mepilex Border Post-Op for post-operative wounds when used according to clinical practice, by assessing dressing wear time from day of surgery to end of dressing use.

The clinical investigation will consist of a retrospective medical record review, which will be completed with data from up to 450 female and male adult subjects who were treated with Mepilex Border Post-Op following elective hip or knee replacement at one clinic in Belgium between January 2016 and February 2021. The data collected for each subject will include those generated in relation to the surgery itself as well as the pre- and post-surgery phases. There is no available data for subjects treated with an alternative to Mepilex Border Post-Op to use as a control group, however, the pre-surgery data will serve as control for some endpoints.

The treatment the subjects received at the clinic included pre-surgery visits, the surgery itself, a short in-patient stay following surgery, and post-surgery follow-up visits at approximately 14 days, 1.5 months, 3 months, 6 months, and 1 year. In addition, the subjects used the commercially available mobile health application moveUP Therapy to support their rehabilitation. The subjects' rehabilitation was tracked and aided with moveUP Therapy as it allows (1) subjects to answer a number of questionnaires; (2) subjects to communicate with their surgeon and physical therapist via a chat function in the app; and (3) subject-specific log entries by the surgeon and physical therapist. The data to be used in this retrospective investigation will be extracted exclusively from moveUP Therapy.

Eligible subjects/medical records will be identified by site personnel through screening moveUP Therapy. Only data from subjects who have consented to the use of their data related to the surgery in an anonymous way for medical research and scientific publications will be extracted.

The investigational device, Mepilex Border Post-Op, was applied as part of the surgery. In the rare event that a dressing change would be required, the subjects were provided with spare dressings and instructions for how to do the change by the treating surgeon or clinic nurse. These instructions included only changing the dressing once at least three corners of the dressing were stained with blood, and to consult the treating surgeon or clinic nurse by sending a moveUP Therapy chat message with a picture of the dressing requesting advice on whether to change or not.

Dressing wear time will be derived from up to three sources:

1. how frequently the subjects have answered the question "Is the dressing dry?" with "Yes, it was changed today";
2. review of potential Health Care Professional log entries for evidence of dressing change(s); and
3. review of potential moveUP Therapy chat messages, including photographs, for evidence of dressing change(s).

Total number of dressings per subject will be derived from the same information as dressing wear time.

ELIGIBILITY:
Inclusion Criteria:

1. Underwent elective knee or hip surgery between January 2016 and February 2021 at the Medisch Centrum Latem, Belgium.
2. Post-operative wound treated with Mepilex Border Post-Op
3. Documented consent in moveUP Therapy
4. Documented consent at Medisch Centrum Latem during pre-op consultation

Exclusion Criteria:

1. Subject missing all answers to the moveUP Therapy question "Is the dressing dry?"

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects/medical records will be identified from a population of adults patients who have had elective hip or knee replacement surgery at the Medisch Centrum Latem, Belgium.
Sampling Method: Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Dressing wear time | From day of surgery to end of dressing use (up to one month)
  Dressing wear time from day of surgery to end of dressing use

SECONDARY OUTCOMES:
Total number of dressings per subject | From day of surgery to end of dressing use (up to one month)
  Total number of dressings/subject from day of surgery to end of dressing use
Time to dressing strikethrough | From day of surgery to end of dressing use (up to one month)
  Time to dressing strikethrough from day of surgery to end of dressing use
Change in physical activity level | Pre-surgery to end of dressing use (up to one month)
  Percentage and absolute change in physical activity level (daily step count) pre-surgery to end of dressing use
Change in the EQ-5D | Pre-surgery to day 83 post surgery
  Percentage and absolute change in the EQ-5D results pre-surgery to day 83.
Change in KOOS or HOOS pain subscale score | pre-surgery to day 42 and day 83 post surgery
  Percentage and absolute change in the KOOS or HOOS pain subscale score pre-surgery to day 42 and day 83
Change in KOOS or HOOS symptoms subscale score | pre-surgery to day 42 and day 83 post surgery
  Percentage and absolute change in the KOOS or HOOS symptoms subscale score pre-surgery to day 42 and day 83
Change in KOOS or HOOS activities of daily living subscale score | pre-surgery to day 42 and day 83 post surgery
  Percentage and absolute change in the KOOS or HOOS activities of daily living subscale score pre-surgery to day 42 and day 83
Change in KOOS or HOOS sport and recreation function subscale score | pre-surgery to day 42 and day 83 post surgery
  Percentage and absolute change in the KOOS or HOOS sport and recreation function subscale score pre-surgery to day 42 and day 83
Change in KOOS or HOOS joint-related quality of life subscale score | pre-surgery to day 42 and day 83 post surgery
  Percentage and absolute change in the KOOS or HOOS joint-related quality of life subscale score pre-surgery to day 42 and day 83
Dressing showerability | From day of surgery to end of dressing use (up to one month)
  Number of incidences (percentage and absolute) of dressing detachment due to subject showering or using water in other ways for personal hygiene reasons

CONTACTS AND LOCATIONS:
Locations (1):
- Medisch Centrum Latem, Sint-Martens-Latem, Belgium